CLINICAL TRIAL: NCT05782673
Title: Assessment of Motor Development With a Wearable in Rural and Low-income Settings: Feasibility and Validity of MAIJU Jumpsuit in Malawi
Brief Title: Assessment of Motor Development With a Wearable in Rural and Low-income Settings
Acronym: MaMa
Status: Active, not recruiting | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Tampere University (Other); University of Helsinki (Other); Kamuzu University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sampsa Vanhatalo, professor in physiology, consultant in clinical neurophysiology, Helsinki University Central Hospital
Other Study IDs: MaMa2022
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Infant Development
Keywords: wearable; motor development; neurodevelopment; child neurology; neurophysiology; activity tracking; developmental assessment; neurological assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: wearable MAIJU for motor assessment — The novel multisensor wearable MAIJU will be used to measure infants' motor performance at home. The recordings are repeated at 2 months intervals betveen 6 and 18 months of age.

SUMMARY:
The MaMa study aims to assess feasibility and validity of an infant wearable in a rural settings. Altogether N~100 infants will be recruited and measured multiple times at homes from age 6 months to age 18 months. Neurodevelopment of the infants is assessed at 18-24 months of age to compare motor development trajectories with the later neurodevelopmental outcome.

DETAILED DESCRIPTION:
The MaMa study aims to assess the feasibility and validity of an infant wearable method to study young infants' neuromotor development in a low income setting. In this method, infants' motor abilities (e.g. variety of different postures and movement types) are measured using a playsuit equipped with movement sensors while the infant is freely playing in his/her native environment, such as home. The data recorded with the wearable sensors is analysed afterwards using an algorithm that quantifies individual movement and posture components as well as delivers holistic interpretations of infant's motor maturity. This method is developed in University of Helsinki, and it is already successfully used in clinical research projects in Finland, Denmark, Italy and USA. Use of movement sensors is common in other wellness and health applications, however wearables of this kind have not been used before for infant's neuromotor assessment. The solution has the advantage that it provides a fully objective and quantified representation of infant's motor activity in his/her native environment; which is not achievable with any of the currently used clinical assessment methods that are typically performed in the outpatient clinic environment.

The study will be conducted in rural Malawi, is East Africa. The investigators will assess the feasibility of the wearable method in a resource poor setting by running a pilot study on approximately five-to-seven-month-old infants. In the first phase, the investigators will assess technical suitability of wearable methods in 20 typically developing infants in the rural settings, and compare the results to those obtained from infants of the same age in Finland. In the second phase, the study will continue as a longitudinal follow-up of these infants and recruit a larger study group of Malawian infants (up to a total N~100), all of whom will undergo repeated assessment with the wearable method, every 6 weeks until the age of 18 months, or until they walk fluently. The results will support constructing motor growth charts for the Malawian infant population. At the age of 24 months, children's neuropsychological performance will be assessed using an assessment battery that was recently adapted for Malawian context; this will allow us to study how early motor development associates with later neurocognitive developmental profile.

There are three potential benefits from performing the study. First, to establish the practical feasibility and utility of a novel method for out-of-hospital neurological assessment in infants. Second, the project will establish functional motor growth charts for Malawian population to serve as a benchmark in any future intervention trial in comparable environments; these can be also compared to data from Finland. Finally, the project will allow assessing links between early motor and later cognitive development, a question with significant global health implications in all cultures.

ELIGIBILITY:
Inclusion Criteria:

* A documented birth date
* Birth at about term age, i.e. between 35 and 42 gestation weeks
* Mother's ability to speak fluently Chi-Chewa, Chi-Yao or English
* Permanent resident of Lungwena Health Centre catchment area
* Availability and willingness of the mother and infant during the period of the study
* Signed or thumb-printed informed consent by the caregiver of the infant

Exclusion Criteria:

* Very early birth (at 7th month or earlier) based on mother's information
* Infant's congenital malformation or severe illness as judged clinically by a study nurse

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants born in the catchment area of Lungwena health center are screened, and the infants are contacted if they fullfil the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor maturation level (BIMS) | The primary outcome BIMS is the level reached by 18 months of age
  BIMS (Baba Infant Motility Score) is a score that combines all recorded postures and movement activities to a holistic estimate of infant's motor maturation. BIMS has a scale from 0 to 100, with higher number being better.

SECONDARY OUTCOMES:
Kilifi Developmental Inventory (KDI) score | 24 months of age
  KDI is a questionnaire based assessment of infants' neurocognitive development at 12-24 months of age. It is validated in the Malawi context. The scale is 0-70, with higher number being better.

CONTACTS AND LOCATIONS:
Overall Officials: Sampsa Vanhatalo, MD PhD, Principal Investigator — professor in physiology, consultant in clinical neurophysiology
Locations (4):
- Finland (2):
  - University of Helsinki, Helsinki
  - BABA, Clinical Trial Unit, New Children's Hospital, Helsinki
- Malawi (2):
  - Lungwena Health Center, Mangochi, Mangochi district
  - Kamuzu University of Health Sciences, Blantyre

IPD SHARING:
Plan to Share IPD: No
data will contain sensitive information that is not allowed to share without additional permission and contracts between relevant insitutions

REFERENCES:
- [Background] Airaksinen M, Gallen A, Kivi A, Vijayakrishnan P, Hayrinen T, Ilen E, Rasanen O, Haataja LM, Vanhatalo S. Intelligent wearable allows out-of-the-lab tracking of developing motor abilities in infants. Commun Med (Lond). 2022 Jun 15;2:69. doi: 10.1038/s43856-022-00131-6. eCollection 2022. PMID 35721830
- [Background] Airaksinen M, Rasanen O, Ilen E, Hayrinen T, Kivi A, Marchi V, Gallen A, Blom S, Varhe A, Kaartinen N, Haataja L, Vanhatalo S. Automatic Posture and Movement Tracking of Infants with Wearable Movement Sensors. Sci Rep. 2020 Jan 13;10(1):169. doi: 10.1038/s41598-019-56862-5. PMID 31932616
- See also: link to presentation of the MAIJU wearable — https://www.babacenter.fi/en.php?k=221282